CLINICAL TRIAL: NCT05591911
Title: Urine Gene Analysis for Pathogen Detection, and Resistance Gene Identification for the Urinary Tract Infection Diagnosis
Brief Title: Urine Gene Analysis for Pathogen Detection
Status: Completed | Type: Observational
Sponsor: David Sheyn (Other)
Collaborators: Vikor Scientific (Unknown); Thermo Fisher Scientific, Inc (Industry)
Responsible Party: Sponsor-Investigator, David Sheyn, Associate Professor, University Hospitals Cleveland Medical Center
Organization: University Hospitals Cleveland Medical Center (Other)
Other Study IDs: STUDY20220767
Record Dates: First submitted 2022-10-19; First posted 2022-10-24 (Actual); Last update posted 2024-10-24 (Actual); Status verified 2024-10

CONDITIONS: Urinary Tract Infections
Keywords: Urinary tract infection; Urine culture; Bacteriel growth; Antibiotics; PCR
MeSH Terms: conditions — Urinary Tract Infections

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: Yes

GROUPS / COHORTS (1):
- Patients over 60 years old presenting with acute urinary tract infection symptoms
  Interventions: Diagnostic Test: Urine PCR testing

INTERVENTIONS:
Diagnostic Test: Urine PCR testing — The urine PCR panel will be performed to evaluate the bacterial growth in the patient's urine who is admitted with acute urinary tract symptoms.

SUMMARY:
The objective of this study is the detection, quantification, and resistance gene identification of pathogens by using the urine of patients with urinary tract infection (UTI) symptoms.

ELIGIBILITY:
Inclusion Criteria:

* Adult men and women 60 years and older who have urinary tract infection
* Can participate in the informed consent process
* Presenting to the clinic with symptoms of UTI or cystitis with no recent history of UTI within the past 21 days
* Able to provide sufficient urine sample volume via clean catch or catheterization for urinalysis, conventional urine culture, and PCR
* Understand and are willing to comply with the study requirements.
* Sample collection able to be sent out the same day via courier

Exclusion Criteria:

* Individuals under 60 years of age
* Unable to provide informed consent
* Urinary diversion of any type
* Chronic indwelling urinary catheter
* No recent history of UTI within the past 21 days
* No antibiotic therapy within the past 21 days
* No recent therapy with Phenazopyridine

Min Age: 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Female and male patients over 60 years old who admit with acute urinary tract infection symptoms to the ambulatory clinics will be included in this research.
Sampling Method: Non-Probability Sample
Enrollment: 96 (Actual)
Dates: Start 2023-06-25 (Actual); Primary Completion 2024-08-31 (Actual); Study Completion 2024-08-31 (Actual)

PRIMARY OUTCOMES:
Time in hours from patient presentation to optimal antibiotic prescription | Up to 30 days
  Time in hours from patient presentation to optimal antibiotic prescription will be evaluated both for urine culture and urine PCR panel utilization.

SECONDARY OUTCOMES:
Antibiotic costs as measured by prescription records | Up to 30 days
  Antibiotic costs spent for UTI treatment will be calculated.
Number of patients with antibiotic change as measured by prescription records | Up to 30 days
  In cases where the UTI cannot be treated with the first antibiotic, other antibiotics used for this purpose will be recorded.
Duration of antibiotic usage as measured by prescription records | Up to 30 days
  Antibiotic usage duration will be recorded.
Number of any HCP visits for same issue as measured by patients reports/medical records | Up to 30 days
  Any visit to HCP for the same issue will be evaluated
Number of hospitalization related to UTI as measured by patients reports/medical records | Up to 30 days
  Hospitalization related to UTI will be recorded.
Number of additional diagnostic procedures completed in relation to UTI as measured by patients reports/medical records | Up to 30 days
  Additional diagnostic procedures completed in relation to UTI will be recorded.

CONTACTS AND LOCATIONS:
Overall Officials: David Sheyn, MD, Principal Investigator — University Hospitals Cleveland Medical Center
Locations (1):
- University Hospitals, Cleveland, Ohio, United States

IPD SHARING:
Plan to Share IPD: No